CLINICAL TRIAL: NCT03769415
Title: HARMONY: Harnessing the Analysis of RNA Expression and Molecular Subtype to Optimize Novel TherapY for Metastatic Breast Cancer
Brief Title: Harnessing Analysis RNA Expression and Molecular Subtype to Optimize Novel TherapY MBCA
Acronym: HARMONY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Veracyte, Inc. (Industry); Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1829
Record Dates: First submitted 2018-11-29; First posted 2018-12-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intrinsic subtyping of Primary Breast Cancer (Experimental): Intrinsic subtype of primary breast tissue from metastatic breast cancer subject will be determined
  Interventions: Device: Intrinsic Subtyping of Primary Breast Cancer

INTERVENTIONS:
Device: Intrinsic Subtyping of Primary Breast Cancer — Primary breast tissue will be sent for Nanostring PAM50 Testing to determine intrinsic subtype

SUMMARY:
The HARMONY trial is an interventional trial enrolling metastatic breast cancer (MBC). Current treatment of breast cancer uses clinical subtype information (e.g. hormone receptor-positive (HR+)) to help guide treatment options. Breast cancer can also be characterized by molecular subtype, but it is not known if this information is helpful in determining treatment when breast cancer has become metastatic. HARMONY will give the treating physician of each participant the molecular subtype of the tumor based on PAM50 testing. The usefulness of this information will be determined through the physician survey. Finding out the molecular subtype of each tumor also allows the investigators to determine if the molecular subtype is different from what is expected based on the clinical subtype. This study will help determine how new types of information about tumors can help choose treatments for MBC

DETAILED DESCRIPTION:
Primary Objectives:

1. To determine if clinical: molecular subtypes differ from expected results 15% of the time
2. To determine if molecular information alters treatment plans, as perceived by treating physicians through the survey.

Subjects will be consented to the trial and archival tissue from the primary tumor will be obtained. Stored tissue from metastatic sites will also be obtained. The physician will be asked what the preferred medications are for the next two lines of treatment. PAM50 testing to determine molecular subtypes will be determined on primary and metastatic tissue. The molecular subtype results of the primary tissue will be returned to the physician, and the physician will again be asked the preferred medications for the next two lines of treatment. The number of times these medications change between the first and second surveys will be determined.

Subjects' active participation will only last as long as the consent process.

ELIGIBILITY:
Inclusion Criteria:

* Women or men at least 18 years of age
* Pathologically documented diagnosis of measurable or evaluable metastatic breast cancer with known ER, PR, and HER2 status determined by the local laboratory on the primary tumor.
* Enrolled before or during first line of treatment for metastatic breast cancer. No more than 1 prior line of therapy in the metastatic setting.
* Accessible medical records for all treatment and response data in the metastatic setting.
* Willing and able to receive medical treatment or follow up by investigators at UNC-Chapel Hill.
* Receiving treatment for metastatic breast cancer.
* Treating physician considers patient well enough for standard of care therapy including chemotherapy.
* Willing to give blood for research purposes upon study enrollment and at first disease progression.
* Available archival primary tumor suitable for molecular analysis. If the primary is not available, willingness to obtain extra samples for research during planned standard of care biopsy, or willingness to undergo biopsy for repeat clinical receptors and molecular analyses.
* Archival metastatic sample available and suitable for molecular analysis. If not available, willingness to undergo biopsy for repeat clinical receptors and molecular analyses. If no archival metastatic sample is available and the metastasis is not amenable to biopsy per treating physician the patient may still be enrolled.
* Be willing and capable of providing informed consent, recognize the experimental nature of the trial, and sign the IRB-approved written informed consent documentations

Exclusion Criteria:

* Does not have tissue available or suitable for molecular analysis, or is unwilling to provide tissue for research at the time of a clinically indicated procedure.
* Has dementia, altered mental status, or any psychiatric or co-morbid condition prohibiting the understanding or rending of informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2030-12-15 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
Change of treatment plan based on physician survey | 4 years
  Number of times physicians change response to the question:" What are the preferred next 2 lines of treatment?" after knowledge of molecular subtype
Overall rate of clinical:molecular primary tumor subtype incongruence | 4 years
  Number of times RNA-based molecular subtype differs from clinically determined subtype in primary breast tumors

SECONDARY OUTCOMES:
Intra-patient PFS ratio comparison | 4 years
  Number of days between initiation of therapy for each line and the date of progression or death (PFS) with adjustment for the expected PFS deterioration over lines of therapy
Intra-patient PFS ratio separated by clinical subtype | 4 years
  Number of days between initiation of therapy for each line and the date of progression or death (PFS) with adjustment for the expected PFS deterioration over lines of therapy separated by each of the follow clinical subtypes: or HR+/HER2-, HR-/HER2+, HR+/HER2+ and HR-/HER2-
Number of patients with HR+/HER2- MBC receiving endocrine therapy on each line of therapy | 4 years
  Number of patients with HR+/HER2- MBC receiving endocrine therapy based on medical record
Rate of molecular discordance | 4 year
  Number of times molecular subtypes determined from primary tissue and molecular subtype determine from metastatic tissue are different
PFS comparison in concordant therapy | 4 years
  PFS for patients receiving clinically-concordant therapy .
PFS comparison in disconcordant therapy | 4 years
  PFS for patients receiving clinically-discordant therapy in congruent tumors

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Carey, MD, FASCO, ScM, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials